CLINICAL TRIAL: NCT02790866
Title: Development and Feasibility Testing of a Lung Cancer Screening Decision Aid
Acronym: LuCaS-DA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Studts (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor-Investigator, Jamie Studts, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 15-0001-P1H
Record Dates: First submitted 2016-05-16; First posted 2016-06-06 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Lung Neoplasms
Keywords: Decision Aid; Informed Decision Making; Shared Decision making; Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LuCaS Decision Aid (Experimental): Access to LuCaS, a web-based lung cancer screening decision aid
  Interventions: Behavioral: LuCaS Decision Aid
- NCI Website (Active Comparator): Access to NCI website on lung cancer screening
  Interventions: Behavioral: NCI Website

INTERVENTIONS:
Behavioral: LuCaS Decision Aid — Web-based Lung Cancer Screening Decision Aid
  Arms: LuCaS Decision Aid
Behavioral: NCI Website — NCI Website on Lung Cancer Screening
  Arms: NCI Website

SUMMARY:
This study evaluates the feasibility and acceptability of LuCaS Choices, a web-based decision aid designed to facilitate informed decision making about participation in lung cancer screening among individuals at high risk of lung cancer due to heavy cigarette smoking.

DETAILED DESCRIPTION:
The proposed project will develop an innovative web-based decision aid (DA) to improve decision making for lung cancer screening (LCS) among individuals at high risk for lung cancer due to cigarette smoking. Recent National Lung Screening Trial (NLST) data demonstrated a 20% relative reduction in lung cancer mortality for low dose computed tomography screening as compared to chest X-ray among individuals at high lung cancer risk. Given that lung cancer is the leading cause of cancer death in the United States with an estimated 160,340 deaths predicted for 2012, the new data have reinvigorated interest in LCS. However, LCS carries substantial risks including a high false positive rate, over-diagnosis, adverse psychosocial consequences, and increased radiation exposure. Further, it is unknown whether LCS would reduce lung cancer mortality among individuals who smoke but do not meet NLST eligibility criteria. Therefore, there is currently no clear best choice for whether a given individual should be screened or not. Decisions about participating in LCS should be well informed and consistent with individual preferences. However, previous data indicate that individuals who do undergo LCS rarely have a thorough understanding of the risks or benefits.

To address this rapidly emerging public health challenge, this research has developed a web-based decision aid (DA) to facilitate informed decision making regarding LCS in individuals at high risk for lung cancer (i.e., cigarette smokers), and will assess feasibility of DA administration and proposed methods for conducting a future randomized clinical trial (RCT) of DA effectiveness. The content of the DA will be based on the investigators previous studies exploring LCS decision making and other recent research.

The specific aim of the currently proposed research are to conduct a feasibility trial of the DA among individuals at high risk of lung cancer due to heavy cigarette smoking. Investigators will recruit participants to assess feasibility of: 1) delivering the DA intervention in a community setting, and 2) conducting research procedures and assessment tools as planned for a future RCT.

ELIGIBILITY:
Inclusion Criteria:

* be at least 40 years of age
* history of 20 or more pack years of smoking
* ability to read and understand English
* must have a personal phone
* must have Internet access

Exclusion Criteria:

* reporting or demonstrating significant psychological distress

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Access Rate POST | Two Weeks (POST)
  Percentage of participants who access LuCaS Choices or National Cancer Institute (NCI) website
Recommendation Rate POST | Two Weeks (POST)
  Percentage of participants who would recommend LuCaS Choices or National Cancer Institute (NCI) website to others who want to learn more about lung cancer screening
Satisfaction Rate POST | Two Weeks (POST)
  Percentage of participants who indicated they were satisfied with LuCaS Choices or National Cancer Institute (NCI) website
Continued Access Rate POST | Two Weeks (POST)
  Percentage of participants who wish to have continued access to LuCaS Choices or National Cancer Institute (NCI) website
Retention Rate POST | Two Weeks (POST)
  Percentage of participants who complete the POST survey
Retention Rate FOL | Four Months (FOL)
  Percentage of participants who complete the FOL survey

SECONDARY OUTCOMES:
Recommendation Rate FOL | Four Months (FOL)
  Percentage of participants who would recommend LuCaS Choices or National Cancer Institute (NCI) website to others who want to learn more about lung cancer screening
Satisfaction Rate FOL | Four Months (FOL)
  Percentage of participants who indicated they were satisfied with LuCaS Choices or National Cancer Institute (NCI) website
Continued Access Rate FOL | Four Months (FOL)
  Percentage of participants who wish to have continued access to LuCaS Choices or National Cancer Institute (NCI) website
Access Rate FOL | Four Months (FOL)
  Percentage of participants who access LuCaS Choices or National Cancer Institute (NCI) website

OTHER OUTCOMES:
Contact Rate | Weekly from study initiation through 12 weeks
  Number of individuals who make email or telephone contact to inquire about the study per week
Eligibility Rate | Weekly from study initiation through 12 weeks
  Number of individuals who are determined to be study eligible
Accrual Rate | Weekly from study initiation through 12 weeks
  Number of individuals who provide informed consent per week

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Studts, PhD, Principal Investigator — University of Kentucky; Margaret M Byrne, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami (FL), Miami, Florida
  - University of Kentucky, Lexington, Kentucky